CLINICAL TRIAL: NCT01269060
Title: Phase 2 Study of Efficacy of Single Incision (Embryonic NOTES) Laparoscopic Colorectal Surgery
Brief Title: Efficacy of Single Incision (Embryonic NOTES) Laparoscopic Colorectal Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Ji Won Park, Principal Investigator, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-484
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer, laparoscopic surgery
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single incision sigmoidectomy (Experimental): Single incision laparoscopic sigmoidectomy for sigmoid colon cancer
  Interventions: Procedure: Single Incision Laparoscopic Surgery

INTERVENTIONS:
Procedure: Single Incision Laparoscopic Surgery — Single Incision Laparoscopic Sigmoidectomy
  Other Names: Embryonic NOTES Sigmoidectomy

SUMMARY:
Laparoscopic colon surgery has been performed widely. As a minimal invasive approach, single incision (Embryonic NOTES) colon surgery has been attempted.

However, there are not sufficient evidences for single incision colon surgery in colon cancer.

The investigators are researching the efficacy and safety of single incision laparoscopic sigmoidectomy in sigmoid colon cancer.

DETAILED DESCRIPTION:
After several randomized clinical trials, laparoscopic colon surgery has been performed widely. As a minimal invasive approach, single Incision (Embryonic NOTES) colon surgery has been attempted. Several studies reported the feasibility of single incision colon surgery.However, there are not sufficient evidences for single incision colon surgery, especially in colon cancer.

The investigators are researching the efficacy and safety of single incision laparoscopic sigmoidectomy in sigmoid colon cancer. Harvested numbers of lymph node will be assessed for the efficacy and postoperative morbidity and mortality will be assess for the safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients should sign a written informed consent
* Age between 18-80
* Patients have sigmoid colon cancer that was proved by pathology
* Adequate bone marrow function Hb ≥ 10g/dl (after treatment for simple iron deficiency anemia) WBC ≥ 3,000/mm3 PLT ≥ 100,000/mm3
* Adequate kidney function Creatinine ≤ 1.5 mg/dl
* No remarkable evidence of heart dysfunction and lung dysfunction

Exclusion Criteria:

* Distant metastasis
* Tumor diameter > 5 cm
* Other organ invasion
* Intestinal obstruction and stent insertion status
* Patient was used steroid
* Patients undergo emergency surgery with multiple symptoms
* Other organ cancer history (except who had radical excision for skin cancer)
* Presence of other serious disease
* Mentally ill patients
* Legally unable to participate in clinical trial
* Lactating or pregnant women
* Patients who will obviously fail to regular follow-up visit or will be off study voluntarily
* Not eligible to participate for other reasons by doctor's decision

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Harvested numbers of lymph node | Within the first 7 days (plus or minus 3 days) after surgery

SECONDARY OUTCOMES:
Postoperative mortality, morbidity | Within 30 days after operation

CONTACTS AND LOCATIONS:
Overall Officials: Jae Hwan Oh, Dr. PhD., Study Chair — Center for Colorectal Cancer, National Cancer Center Korea
Locations (1):
- National Cancer Center Hospital, Goyang-si, Gyeonggi-do, South Korea